CLINICAL TRIAL: NCT02900651
Title: A Phase I/II, Multicenter, Open-label Study of MAK683 in Adult Patients With Advanced Malignancies
Brief Title: Safety and Efficacy of MAK683 in Adult Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision of early termination was made due to business reasons, and was not based on any safety or tolerability concerns for MAK683
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMAK683X2101; 2016-001860-12 (EudraCT Number)
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: MAK683, DLBCL, EED - Embryonic ectoderm development, EZH2 - Enhancer of zeste homolog 2
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I - All (Experimental): advanced stage (relapsed/refractory or recurrent/metastatic) malignancy limited to the following malignancies; DLBCL, nasopharyngeal carcinoma, gastric cancer, ovarian cancer, prostate cancer and sarcoma.
  Interventions: Drug: MAK683

INTERVENTIONS:
Drug: MAK683 — Drug: MAK683

SUMMARY:
The purpose of this Phase I/II study is to establish the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) and to evaluate the safety, antitumor activity and pharmacokinetic (PK) profile of MAK683 in patients with advanced malignancies such as Diffuse Large B cell Lymphoma (DLBCL), nasopharyngeal carcinoma (NPC) or other advanced solid tumors for whom no further effective standard treatment is available.

DETAILED DESCRIPTION:
The purpose phase I of this trial is to characterize safety and tolerability and determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of MAK683.

The purpose of the phase II of this trial is to evaluate the anti-tumor activity of MAK683. Phase II part will not be opened.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG): 0 to 2
2. Relapsed or refractory diffuse large B cell lymphoma with measurable disease as determined by Non-Hodgkin's Lymphoma Cheson response criteria (2014)
3. Advanced or recurrent/metastatic solid tumor, including nasopharyngeal carcinoma, castration-resistant prostate cancer, gastric cancer, ovarian clear cell carcinoma and sarcoma, with measurable disease as determined by RECIST 1.1.

Exclusion Criteria:

1. Other malignant diseases than the ones being treated in this study
2. Severe and/or uncontrolled medical conditions that in the investigator's opinion could affect the safety of individual or impair the assessment of study result.
3. B-cell lymphoma patients who have received prior allogeneic stem cell transplant
4. Patient have received anti-cancer therapies within defined time frames prior to the first dose of study treatment
5. Symptomatic central nervous system (CNS) involvement which are neurologically unstable or requiring increasing doses of steroids to control.
6. Patient having out of range laboratory values defined as:

1) Insufficient bone marrow function at screening:

* Platelets ≤ 50,000/mm3
* Hemoglobin (Hgb) ≤ 80 g/L
* Absolute neutrophil count (ANC) ≤ 1000/mm3 2) Insufficient hepatic and renal function at screening:
* ALP, ALT, and AST > 3 x ULN (>5 x ULN if subject has liver metastases)
* Total bilirubin >1.5 x ULN
* Serum creatinine > 1.5 x ULN and/or creatinine clearance ≤ 50 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | up to 28 days
  Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Safety and tolerability | up to approximately 3 years
  Incidence and severity of AEs, SAEs, changes in laboratory values, vital signs and ECGs, dose interruptions and reductions

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 30 months
Duration of overall response (DOR) | up to 30 months
Progression-free survival (PFS) | up to 30 months
Best Overall Response (BOR) | up to 30 months
Peak Plasma Concentration (Cmax) of MAK683 | 30 months
  Pharmacokinetic profile of MAK683
Area Under the Plasma Concentration (AUC) Time Curve of MAK683 | 30 months
  Pharmacokinetic profile of MAK683
Half-Life of MAK683 | 30 months
  Pharmacokinetic profile of MAK683
H3K27 tri methylation level in PBMC | up to day 15
  Cycle 1 Day 1,8,15 Cycle 2 Day1 Cycle 3 Day 1 End of treatment (EOT); Disease progression PBMC: peripheral blood mononuclear cell

CONTACTS AND LOCATIONS:
Locations (16):
- United States (3):
  - UCSF ., San Francisco, California
  - UCLA Santa Monica Hematology Oncology, Santa Monica, California
  - Uni Of TX MD Anderson Cancer Cntr Dept of Onc, Houston, Texas
- Novartis Investigative Site, Toronto, Ontario, Canada
- China (2):
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Villejuif, France
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Freiburg im Breisgau
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Japan (2):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sunto Gun, Shizuoka
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ribrag V, Iglesias L, De Braud F, Ma B, Yokota T, Zander T, Spreafico A, Subbiah V, Illert AL, Tan D, Santoro A, Munster PN, Suehiro Y, Wang Y, Ji DM, Chen S, Beltz K, Suenaga N, Ramkumar T, Luo F, Lai C, Wainberg ZA. A first-in-human phase 1/2 dose-escalation study of MAK683 (EED inhibitor) in patients with advanced malignancies. Eur J Cancer. 2025 Feb 5;216:115122. doi: 10.1016/j.ejca.2024.115122. Epub 2024 Nov 16. PMID 39793445
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18338